CLINICAL TRIAL: NCT00136019
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel Group Trial to Investigate the Efficacy and Safety of SPM 927 (400mg/Day and 600mg/Day) as Adjunctive Therapy in Subjects With Partial Seizures With or Without Secondary Generalization
Brief Title: SPM 927 (400mg/Day and 600mg/Day) as Adjunctive Therapy in Subjects With Partial Seizures With or Without Secondary Generalization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0754
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2010-07

CONDITIONS: Epilepsy
Keywords: Epilepsy with partial seizures
MeSH Terms: conditions — Epilepsy | interventions — 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-

INTERVENTIONS:
Drug: SPM 927

SUMMARY:
Male and female patients between 16 and 70 years of age who are diagnosed with epilepsy with partial seizures and are taking up to 3 medications for this medical condition will take part in a research study at approximately 85 different locations in the United States.

The purpose of the study is to evaluate the effectiveness, safety and tolerability of consistent dosages of a study drug (lacosamide [SPM 927]) taken orally twice a day for about five months.

Each patient who qualifies and chooses to participate in the study will receive placebo (inactive drug) or gradually increasing doses of lacosamide up to the target dose of 400mg/day or 600mg/day. The target dose or placebo will be maintained for 12 weeks.

The study clinic visits will include a medical history and physical exam, electrocardiogram (ECG), blood and urine sample collection, and completion of a seizure diary.

Patients who complete the study may enroll in an extension trial and receive active study drug.

ELIGIBILITY:
Inclusion Criteria:

* Epilepsy with partial seizures

Exclusion Criteria:

* Subject received SPM 927 in a previous trial

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2004-03; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Efficacy is evaluated based on reduction in seizure frequency, 50 percent reduction in seizures, number and percentage of seizure-free days, and achievement of seizure-free status.

SECONDARY OUTCOMES:
Safety of lacosamide was evaluated with the monitoring of adverse events (AEs), ECGs, vital signs, and clinical laboratory data.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma

REFERENCES:
- [Result] Chung S, Sperling MR, Biton V, Krauss G, Hebert D, Rudd GD, Doty P; SP754 Study Group. Lacosamide as adjunctive therapy for partial-onset seizures: a randomized controlled trial. Epilepsia. 2010 Jun;51(6):958-67. doi: 10.1111/j.1528-1167.2009.02496.x. Epub 2010 Jan 27. PMID 20132285
- [Result] Sake JK, Hebert D, Isojarvi J, Doty P, De Backer M, Davies K, Eggert-Formella A, Zackheim J. A pooled analysis of lacosamide clinical trial data grouped by mechanism of action of concomitant antiepileptic drugs. CNS Drugs. 2010 Dec;24(12):1055-68. doi: 10.2165/11587550-000000000-00000. PMID 21090839
- [Result] Borghs S, de la Loge C, Cramer JA. Defining minimally important change in QOLIE-31 scores: estimates from three placebo-controlled lacosamide trials in patients with partial-onset seizures. Epilepsy Behav. 2012 Mar;23(3):230-4. doi: 10.1016/j.yebeh.2011.12.023. Epub 2012 Feb 15. PMID 22341962
- [Derived] Biton V, Gil-Nagel A, Isojarvi J, Doty P, Hebert D, Fountain NB. Safety and tolerability of lacosamide as adjunctive therapy for adults with partial-onset seizures: Analysis of data pooled from three randomized, double-blind, placebo-controlled clinical trials. Epilepsy Behav. 2015 Nov;52(Pt A):119-27. doi: 10.1016/j.yebeh.2015.09.006. Epub 2015 Sep 27. PMID 26414341